CLINICAL TRIAL: NCT05831189
Title: A Multi-center, Single-arm Trial Exploring the Safety and Clinical Effectiveness of RBX2660 Administered by Colonoscopy to Adults With Recurrent Clostridioides Difficile Infection
Acronym: CDI-SCOPE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 000416
Record Dates: First submitted 2023-04-14; First posted 2023-04-26 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Clostridium Difficile Infection Recurrence
Keywords: C. Difficile Diarrhea; Clostridium Difficile; CDI; FMT; Fecal Microbiota Transplant; Microbiota Restoration Therapy; Diarrhea; Microbial Suspension; Fecal Transplant; C Difficile Colitis; Clostridium Difficile Associated Diarrhea; C diff diarrhea; C Difficile; C diff
MeSH Terms: conditions — Diarrhea; Enterocolitis, Pseudomembranous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- RBX2660 (Experimental)
  Interventions: Drug: RBX2660

INTERVENTIONS:
Drug: RBX2660 — RBX2660 should be administered to the right side of the colon (i.e., between the ileocecal valve and the hepatic flexure of the colon).
  Other Names: REBYOTA®

SUMMARY:
This trial will be initiated to explore whether RBX2660 (REBYOTA®) could be suitable for administration by the practice of colonoscopy. More specifically, the purpose of this trial is to explore the safety and clinical effectiveness of RBX2660 when delivered by colonoscopy to adults with rCDI. The experience of physicians will be documented through a physician-experience questionnaire to explore the usability of RBX2660 in clinical practice for colonoscopic administration. Furthermore, to explore the patient-experience of RBX2660 treatment, each trial participant will be offered to undergo a structured interview.

ELIGIBILITY:
Inclusion Criteria:

* have documented evidence of rCDI (≥1 recurrence after a primary CDI episode)
* be undergoing antibiotic treatment for the qualifying rCDI episode that was diagnosed by a stool test for the presence of toxigenic C. difficile or C. difficile toxin
* be eligible for FMT as judged by the investigator or current treatment guidelines for rCDI in the US
* be a candidate for colonoscopy as judged by the investigator

Exclusion Criteria:

* Use or planned use of systemic antibiotics for an indication other than the qualifying rCDI episode.
* Current uncontrolled chronic diarrhea not related to CDI.
* Receipt of CDI vaccine or treatment with CDI monoclonal antibodies within the past 12 months before screening.
* Evidence of active, severe, or fulminant colitis, diagnosis of toxic megacolon or have a current colostomy or ileostomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2023-04-21 (Actual); Primary Completion 2025-01-17 (Actual); Study Completion 2025-01-17 (Actual)

PRIMARY OUTCOMES:
RBX2660-related treatment-emergent adverse events (TEAEs) after RBX2660 treatment delivered by colonoscopy through 8 weeks, or treatment failure | 8 weeks after RBX2660 treatment delivered by colonoscopy

SECONDARY OUTCOMES:
Recurrence of Clostridioides difficile infection (CDI) within 8 weeks after RBX2660 treatment delivered by colonoscopy. | Within 8 weeks after RBX2660 treatment delivered by colonoscopy
Time to CDI recurrence from baseline through 8 weeks after RBX2660 treatment delivered by colonoscopy | 8 weeks after RBX2660 treatment delivered by colonoscopy
Physician-experience, as determined by questionnaire, documenting subjective experience of investigators on usability of RBX2660 in clinical practice when delivered by colonoscopy | At Day 1 (baseline visit)
Physician perception of patient benefit, as determined by Clinician Global Impression of Improvement (CGI-I) at 8 weeks, or at treatment failure, after RBX2660 treatment delivered by colonoscopy | 8 weeks after RBX2660 treatment delivered by colonoscopy
Patient-experience interview at 8 weeks, or at treatment failure, after RBX2660 treatment delivered by colonoscopy | 8 weeks after RBX2660 treatment delivered by colonoscopy
TEAEs, including type, intensity, and causality | Up to 8 weeks after RBX2660 treatment delivered by colonoscopy
Serious adverse events (SAEs) | Up to 8 weeks after RBX2660 treatment delivered by colonoscopy
Adverse events of special interest (AESIs): septic shock, toxic megacolon, colonic perforation, and emergency colectomy | Up to 8 weeks after RBX2660 treatment delivered by colonoscopy
Adverse events leading to death or intensive care unit (ICU) admission | Up to 8 weeks after RBX2660 treatment delivered by colonoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Compliance, Study Director — Ferring Pharmaceuticals
Locations (12):
- United States (12):
  - Ferring Investigational Site, North Little Rock, Arkansas
  - Ferring Investigational Site, Camarillo, California
  - Ferring Investigational Site, Hamden, Connecticut
  - Ferring Investigational Site, Idaho Falls, Idaho
  - Ferring Investigational Site, Gurnee, Illinois
  - Ferring Investigational Site, Shreveport, Louisiana
  - Ferring Investigational Site, Plymouth, Minnesota
  - Ferring Investigational Site, Rochester, Minnesota
  - Ferring Investigational Site, Cleveland, Ohio
  - Ferring Investigational Site, Oklahoma City, Oklahoma
  - Ferring Investigational Site, Burke, Virginia
  - Ferring Investigational Site, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Khanna S, Yoho D, Van Handel D, Clark BJ, Awad T, Guthmueller B, Armandi D, Knapple W, Safdar N, Baggott B, Simon K, Feuerstadt P. Safety and effectiveness of fecal microbiota, live-jslm (REBYOTA(R)) administered by colonoscopy for prevention of recurrent Clostridioides difficile infection: 8-week results from CDI-SCOPE, a single-arm, phase IIIb trial. Therap Adv Gastroenterol. 2025 Apr 22;18:17562848251339697. doi: 10.1177/17562848251339697. eCollection 2025. PMID 40321366
- [Result] Khanna S, Yoho D, Van Handel D, Clark BJ, Awad T, Guthmueller B, Armandi D, Knapple W, Safdar N, Baggott B, Simon K, Feuerstadt P. Prevention of recurrent Clostridioides difficile infection by fecal microbiota, live-jslm (REBYOTA(R)) administered via colonoscopy: 6-month data from the single-arm phase IIIb CDI-SCOPE trial. Therap Adv Gastroenterol. 2025 Nov 9;18:17562848251396744. doi: 10.1177/17562848251396744. eCollection 2025. PMID 41230019
- [Result] McCool-Myers M, Umanzor-Figueroa C, Symonds T, Landeira M, Awad T, Armandi D, Guthmueller B & Khanna S. Patient-reported benefits of colonoscopically administered microbiota restoration therapy: a qualitative study of adult patients with recurrent Clostridioides difficile infection. Therapeutic Advances in Gastroenterology. 2025 Nov 14; 18:17562848251392102. doi: 10.1177/17562848251392102.
- [Derived] McCool-Myers M, Umanzor-Figueroa C, Symonds T, Landeira M, Awad T, Armandi D, Guthmueller B, Khanna S. Patient-reported benefits of colonoscopicallyadministered microbiota restoration therapy: a qualitative study of adult patients with recurrent Clostridioides difficile infection. Therap Adv Gastroenterol. 2025 Nov 14;18:17562848251392102. doi: 10.1177/17562848251392102. eCollection 2025. PMID 41647268
- See also: Safety and effectiveness of fecal microbiota, live-jslm (REBYOTA(R)) administered by colonoscopy for prevention of recurrent Clostridioides difficile infection: 8-week results from CDI-SCOPE, a single-arm, phase IIIb trial — https://pubmed.ncbi.nlm.nih.gov/40321366/
- See also: Prevention of recurrent Clostridioides difficile infection by fecal microbiota, live-jslm (REBYOTA(R)) administered via colonoscopy: 6-month data from the single-arm phase IIIb CDI-SCOPE trial. — https://pubmed.ncbi.nlm.nih.gov/41230019/